CLINICAL TRIAL: NCT05664386
Title: Effect of Ciprofol Infusion for Induction and Maintenance on Hemodynamics and Postoperative Recovery in Patients Undergoing Thoracoscopic Lobectomy : a Randomized, Controlled Trial
Brief Title: Effect of Ciprofol Infusion for Induction and Maintenance on Hemodynamics and Postoperative Recovery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiumei Song (Other)
Responsible Party: Sponsor-Investigator, Xiumei Song, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20221128C
Record Dates: First submitted 2022-11-29; First posted 2022-12-23 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hemodynamics; Postoperative Recovery; Anesthesia
Keywords: Ciprofol; Hemodynamics; Postoperative Recovery; propofol
MeSH Terms: interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): According to grouping，patients were premeditated with injection of Propofol 2-2.5mg / kg IV . If BIS is ≤ 60, Tracheal intubation was facilitated with cisatracurium 0.2mg/kg a IV and sufentanil 0.3 μ g / kg IV. if BIS is >60, propofol 1mg/kg was titrated intravenously, with an interval of more than 1min until the BIS is ≤ 60，and intubation was performed after cisatracurium and sufentanil injected .General anesthesia was maintained with Propofol and remifentanil.Then propofol was maintained in group P at 4-12 mg/kg/h and remifentanil was maintained at 0.1-0.3 ug/kg/min .BIS was kept at 40 ~ 60 during the surgery, and infusion drugs were stopped at the end of the operation. The patients were Transfered to Postanesthesia care unit(PACU) after the operation.
  Interventions: Drug: propofol
- ciprofol group (Experimental): Group C was given ciprofol 0.4 ~ 0.5mg/kg, if bispectral index(BIS) value ≤60 during anesthesia induction, cisatracurium 0.2mg/kg and sufentanil 0.5μg/kg were injected intravenously, endotracheal intubation was performed after the improvement of muscle relaxation. If the BIS value was greater than 60, ciprofol 0.2mg/kg each time, and the interval of administration was greater than 1min, until BIS≤60. Cisatracurium and sufentanil were injected intravenously, followed by endotrachealintubation.Ciprofol was maintained in Group C at 0.8-2.5 mg/kg/h and remifentanil was maintained at 0.1-0.3 ug/kg/min . Intermittent addition of cisatracurium,Sufentanil was added as required, and total dosage of Sufentanil was 0.7ug ~ 1ug/kg. BIS was kept at 40 ~ 60 during the surgery, and infusion drugs were stopped at the end of the operation. The patients were Transfered to Postanesthesia care unit(PACU) after the operation.
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: propofol — propofol 2～2.5mg/kg was used for anesthesia induction. propofol is an intravenous sedative-hypnotic and a short-acting GABAA receptor agonist. It activates GABAergic neurons by enhancing chloride ion influx. It is used for anesthesia of induction and maintenance.
  Arms: propofol group
Drug: ciprofol — Ciprofol 0.4～0.5mg/kg was used for anesthesia induction. Ciprofol is an intravenous sedative-hypnotic and a short-acting GABAA receptor agonist. It activates GABAergic neurons by enhancing chloride ion influx. It is used for anesthetic induction and maintenance agents include rapid induction of general anesthesia, rapid recovery of consciousness, minimal residual effects on the central nervous system and less injection pain.
  Arms: ciprofol group

SUMMARY:
To study the Effect of Ciprofol Infusion for Induction and Maintenance of anesthesia on Hemodynamics and Postoperative Recovery in Patients Undergoing Thoracoscopic Lobectomy:a randomized, controlled trial.

DETAILED DESCRIPTION:
Patients undergoing Thoracoscopic Lobectomy aged 18~65 years old were randomly assigned to Group P and Group C . Group P was given propofol 2 ~ 2.5mg/kg, group C was given ciprofol 0.4 ~ 0.5mg/kg, if bispectral index(BIS) value ≤60 during anesthesia induction, cisatracurium 0.2mg/kg and sufentanil 0.5μg/kg were injected intravenously, endotracheal intubation was performed after the improvement of muscle relaxation. If the BIS value was greater than 60, propofol was added intravenously 1mg/kg each time or ciprofol 0.2mg/kg each time, and the interval of administration was greater than 1min, until BIS≤60. Cisatracurium and sufentanil were injected intravenously, followed by endotracheal intubation.Then propofol was maintained in group P at 4-12 mg/kg/h and remifentanil was maintained at 0.1-0.3 ug/kg/min .Ciprofol was maintained in Group C at 0.8-2.5 mg/kg/h and remifentanil was maintained at 0.1-0.3 ug/kg/min . Intermittent addition of cisatracurium. Sufentanil was added as required, and total dosage of Sufentanil was 0.7ug ~ 1ug/kg. BIS was kept at 40 ~ 60 during the surgery, and infusion drugs were stopped at the end of the operation. The patients were Transfer to Postanesthesia care unit(PACU) after the operation.

The primary outcomes were the fluctuations in hemodynamic parameters during induction and the surgery. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MAP),heart rate (HR) and BIS values at various time points were collected.

The secondary outcome were as follows:

1. The time of lose consciousness（LOC） during the induction, The Time and dosage of additional drug, and the BIS value during the induction process.
2. The incidence of adverse events such as injection pain, body movement, muscle twitching, hypotension, hypertension, bradycardia or tachycardia, cough and bronchospasm during induction.
3. quality of recovery 15（QOR15） score at pre-operation（Preop） 、on the first day of postoperation （POD1）and on the second day of postoperation （POD2） .
4. the recovery time of consciousness (ROC）, extubation time, PACU stay time, postoperative hospital stay time.
5. Incidence of postoperative nausea and vomiting, incidence of postoperative agitation and delayed recovery, and intraoperative awareness.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA)Ⅰ～Ⅱ grade;
* 18-65 years;
* Body mass index (BMI) 20-30kg/m2 ;
* Scheduled for thoracoscopic lobectomy under general anesthesia;

Exclusion Criteria:

* Refused to participate in the clinical study;
* Predictable airway difficulties requiring awake intubation;
* Allergy to the drugs which were used in this study;
* Tracheal intubation failed for twice;
* Patients with mental diseases or consciousness disorder;
* long-term use of sedatives or Antidepressants;
* Patients who are participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic fluctuations: Systolic blood pressure(SBP) | during anesthesia induction，perioperative
  Systolic blood pressure(SBP) during anesthesia induction and surgery.
Hemodynamic fluctuations: Diastolic blood pressure(DBP) | during anesthesia induction，perioperative
  Diastolic blood pressure(DBP) during anesthesia induction and surgery.
Hemodynamic fluctuations: mean blood pressure (MAP) | during anesthesia induction，perioperative
  MAP during anesthesia induction and surgery.
Hemodynamic fluctuations: Heart rate (HR) | during anesthesia induction，perioperative
  Heart rate (HR) during anesthesia induction and surgery.

SECONDARY OUTCOMES:
The time of lose consciousness（LOC） during the induction | during anesthesia induction
  The time of lose consciousness（LOC） during the induction was defined as from the drug was administered until the patients loss of consciousness(when the BIS≤60)
The incidence of adverse events during induction | during induction
  The incidence of adverse events such as injection pain, body movement, muscle twitching, hypotension, hypertension, bradycardia or tachycardia, cough and bronchospasm during induction.
quality of recovery | pre-operation, postoperation of day 1 ,postoperation of day2
  quality of recovery 15（QOR15） score at pre-operation（Preop） 、 postoperation day 1 ,postoperation of day2
postoperative recovery | 2 hours after surgery
  Incidence of postoperative nausea and vomiting was record use Classification of nausea and vomiting
Incidence of intraoperative awareness | 2 hours after surgery
  Brice Questionnaire was used to assess the occurrence of intraoperative awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Xiumei Song, PH.D, Study Chair — Qian fo shan hospitial of shan dong province, China
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload and share data with other researchers. Protecting patient privacy when sharing patient-level data from clinical trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: study protocol and Informed Consent Form will available before 2024/1/1 Statistical Analysis Plan and Clinical Study Report will available before 2024/6/1
Access Criteria: All registered researchers

REFERENCES:
- [Background] Teng Y, Ou M, Wang X, Zhang W, Liu X, Liang Y, Li K, Wang Y, Ouyang W, Weng H, Li J, Yao S, Meng J, Shangguan W, Zuo Y, Zhu T, Liu B, Liu J. Efficacy and safety of ciprofol for the sedation/anesthesia in patients undergoing colonoscopy: Phase IIa and IIb multi-center clinical trials. Eur J Pharm Sci. 2021 Sep 1;164:105904. doi: 10.1016/j.ejps.2021.105904. Epub 2021 Jun 8. PMID 34116176
- [Background] Wang X, Wang X, Liu J, Zuo YX, Zhu QM, Wei XC, Zou XH, Luo AL, Zhang FX, Li YL, Zheng H, Li H, Wang S, Wang DX, Guo QL, Liu CM, Wang YT, Zhu ZQ, Wang GY, Ai YQ, Xu MJ. Effects of ciprofol for the induction of general anesthesia in patients scheduled for elective surgery compared to propofol: a phase 3, multicenter, randomized, double-blind, comparative study. Eur Rev Med Pharmacol Sci. 2022 Mar;26(5):1607-1617. doi: 10.26355/eurrev_202203_28228. PMID 35302207
- [Background] Qin K, Qin WY, Ming SP, Ma XF, Du XK. Effect of ciprofol on induction and maintenance of general anesthesia in patients undergoing kidney transplantation. Eur Rev Med Pharmacol Sci. 2022 Jul;26(14):5063-5071. doi: 10.26355/eurrev_202207_29292. PMID 35916802
- [Background] Chen BZ, Yin XY, Jiang LH, Liu JH, Shi YY, Yuan BY. The efficacy and safety of ciprofol use for the induction of general anesthesia in patients undergoing gynecological surgery: a prospective randomized controlled study. BMC Anesthesiol. 2022 Aug 3;22(1):245. doi: 10.1186/s12871-022-01782-7. PMID 35922771
- [Background] Ding YY, Long YQ, Yang HT, Zhuang K, Ji FH, Peng K. Efficacy and safety of ciprofol for general anaesthesia induction in elderly patients undergoing major noncardiac surgery: A randomised controlled pilot trial. Eur J Anaesthesiol. 2022 Dec 1;39(12):960-963. doi: 10.1097/EJA.0000000000001759. No abstract available. PMID 36214498
- [Derived] Guo N, Cao J, Duan M, Zhou F, Wang W, Xu L, Wei C, Song X. Effects of ciprofol infusion on hemodynamics during induction and maintenance of anesthesia and on postoperative recovery in patients undergoing thoracoscopic lobectomy: Study protocol for a randomized, controlled trial. PLoS One. 2024 Jul 10;19(7):e0305478. doi: 10.1371/journal.pone.0305478. eCollection 2024. PMID 38985796
- See also: Liu J, Wang D , Zuo Y, MI W, Yao S, Yu W. Guidelines on clinical application of ciprofol. Chin J Anesthesiol, 2021,41 (2): 129-132 — http://rs.yiigle.com/CN131073202102/1326216.htm